CLINICAL TRIAL: NCT01755520
Title: A Randomized, Parallel Group, Double-Blind Study of Ticagrelor Compared With Aspirin for Prevention of Vascular Events in Patients Undergoing Coronary Artery Bypass Graft Operation TiCAB- Ticagrelor in CABG
Brief Title: Study Comparing Ticagrelor With Aspirin for Prevention of Vascular Events in Patients Undergoing CABG
Acronym: TiCAB
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DSMB Interim Analyses
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GE IDE No. D00112; 2012-003630-16 (EudraCT Number)
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Coronary Artery Disease; Stable Angina; Acute Coronary Syndrome
Keywords: CABG; CAD; antiplatelet drug; Ticagrelor; Aspirin
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable; Acute Coronary Syndrome | interventions — Ticagrelor; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor (Experimental): Intervention: Drug: Ticagrelor verum + Aspirin placebo
  Interventions: Drug: Ticagrelor; Drug: Placebo - Aspirin
- Aspirin (Active Comparator): Intervention: Drug: Aspirin verum + Ticagrelor placebo
  Interventions: Drug: Aspirin; Drug: Placebo - Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — 90mg twice daily dose
  Other Names: Brilique
  Arms: Ticagrelor
Drug: Aspirin — Aspirin 100mg once daily
  Other Names: ASS
  Arms: Aspirin
Drug: Placebo - Ticagrelor — Placebo
  Other Names: Placebo
  Arms: Aspirin
Drug: Placebo - Aspirin — Placebo
  Other Names: Placebo
  Arms: Ticagrelor

SUMMARY:
The primary objective of this study ist to test the hypothesis that ticagrelor is superior to Aspirin (ASA) fort he prevention of major cardio- and cerebrovascular events (MACCE) in patients undergoing artery bypass operation.

The primary efficiacy MACCE-endpoint is the composite of cardiovascular death, myocardial infarction, recurent revascularisation, and stroke at twelve month after coronary artery bypass operation.

DETAILED DESCRIPTION:
For stable patients who underwent coronary bypass operation, Aspirin alone currently represents the gold standard of antiplatelet treatment.

The CABG substudy of the PLATO-trial (http://www.nejm.org/doi/full/10.1056/NEJMoa0904327) comprising more than 1200 patients has convincingly shown a high significant reduction of cardiovascular and all-cause mortality for patients recieving Aspirin and Ticagrelor as compared to those subjects randomized to Aspirin plus Clopidogrel. Moreover the results of the PLATO CABG substudy showed that benefits of Ticagrelor increase with decreasing Aspirin doses. Therefore Ticagrelor monotherapy (2x 90mg/day) appears to offer the best balance of safety with anticipated improved efficacy over Aspirin (1x 100mg/day) alone, but until now there are no further data available to support this hypothesis.

Hence this study (TiCAB) is assigned as a pivotal efficacy and safety study of Ticagrelor in patients undergoing coronary artery bypass operation and to test the hypothesis that ticagrelor is superior to Aspirin for the prevention of major cardio- and cerebrovascular events (MACCE) in this patient population.

The TiCAB trial is designed as a randomized, double-blind, double-dummy, parallel group, phase III, multicenter study, comparing the efficacy and safety of Ticagrelor 90mg administered twice daily with Aspirin 100mg once daily, for the prevention of MACCE within the first year after CABG operation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older
2. Informed, written consent by the patient
3. Indication for CABG surgery:

   * coronary three vessel disease, or
   * left main stenosis, or
   * two vessel disease with impaired left ventricular function (<50%)

Exclusion Criteria:

1. Cardiogenic shock, haemodynamic instability
2. Indication for oral anticoagulation or dual antiplatelet therapy that can not be stopped after CABG
3. Need for concomitant non-coronary surgery (e.g. valve replacement)
4. Intolerance of or Allergy to Ticagrelor or ASA or any of their ingredients
5. History of bleeding diathesis within three months prior presentation
6. History of significant gastrointestinal bleeding within six months prior presentation
7. History of intracranial hemorrhage
8. History of moderate to severe liver impairment (Child Pugh B or C)
9. Chronic renal insufficiency requiring dialysis
10. Patient with an increased risk of bradycardic events (e.g. patients without a pacemaker who have sick sinus syndrome, 2nd or 3rd degree AV block or bradycardic-related syncope)
11. Known, clinically important thrombocytopenia (i.e. <100.000/µl)
12. Known, clinically important anaemia (i.e. <10mg/dl)
13. Participation in another investigational drug or device study in the last 30 days
14. Pregnancy or lactation (for premenopausal women 2 methods of reliable contraception, one of which must be barrier method, are required); in women with childbearing potential a pregnancy test is mandatory
15. Concomitant oral or intravenous therapy (see examples below) with strong CYP3A inhibitors, CYP3A substrates with narrow therapeutic indices, or strong CYP3A inducers which cannot be stopped for the course of the study

    * Strong inhibitors: ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, over 1 litre daily of grapefruit juice.
    * Substrates with narrow therapeutic index: cyclosporine, quinidine.
    * Strong inducers: rifampin/rifampicin, phenytoin, carbamazepine.
16. Life expectancy less than 12 months that may result in protocol non-compliance or a risk for being lost to follow-up, active cancer
17. Indication for major surgery (e.g. cancer treatment, carotid surgery, cerebral surgery, major vascular surgery)
18. Previous enrollment or randomization of treatment in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1893 (Actual)
Dates: Start 2013-04-24; Primary Completion 2018-05-19 (Actual); Study Completion 2018-05-19 (Actual)

PRIMARY OUTCOMES:
MACCE | at 12 months after coronary artery bypass surgery
  Composite of cardiovascular death, myocardial infarction, target vessel revascularization, and stroke

SECONDARY OUTCOMES:
Cardiovascular death | at 12 months after coronary artery bypass surgery
Major bleeding events | within 12 months after coronary arerty bypass surgery
  Incidence of major bleeding events
All cause death | at 12 months after coronary artery bypass surgery
  All cause death
Myocardial Infarction | at 12 months after coronary artery bypass surgery
Target Lesion Revascularization | at 12 months after coronary artery bypass surgery
Stroke | at 12 months after coronary artery bypass surgery

CONTACTS AND LOCATIONS:
Overall Officials: Heribert Schunkert, MD, Study Chair — Deutsches Herzzentrum Munich Germany
Locations (29):
- Austria (2):
  - Medizinische Universität Wien, Vienna
  - Klinikum Wels-Grieskirchen, Wels
- Germany (26):
  - Deutsches Herzzentrum München, Munich, Bavaria
  - Herzzentrum Brandenburg in Bernau, Bernau bei Berlin, Brandenburg
  - Herz- und Kreislaufzentrum Rothenburg an der Fulda, Rotenburg an der Fulda, Hesse
  - Universitätsklinikum Jena, Jena, Thuringia
  - Universitätsklinikum Aachen, Aachen
  - Herz- und Gefäßzentrum, Bad Bevensen
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Charité Universitätsmedizin Berlin, Berlin
  - Deutsches Herzzentrum Berlin, Berlin
  - Gesundheit Nord gGmbH, Klinikum Links der Weser gGmbH, Bremen
  - Sana Herzzentrum Cottbus GmbH, Cottbus
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - St. Antonius Hospital, Eschweiler
  - Universitäts-Herzzentrum Freiburg / Bad Krozingen, Freiburg im Breisgau
  - Universitätsklinikum Gießen, Giessen
  - Universitätsmedizin Göttingen, Göttingen
  - Asklepios Klinik St.Georg, Hamburg
  - Universitäres Herzzentrum Hamburg GmbH, Hamburg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Herzzentrum Leipzig GmbH, Leipzig
  - Klinikum Ludwigshafen, Ludwigshafen
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Klinikum Nürnberg Süd, Nuremberg
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
- Schweizer Herz- und Gefässchirurgie, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sandner SE, Schunkert H, Kastrati A, Wiedemann D, Misfeld M, Boning A, Tebbe U, Nowak B, Stritzke J, Laufer G, von Scheidt M; TiCAB Investigators. Ticagrelor monotherapy versus aspirin in patients undergoing multiple arterial or single arterial coronary artery bypass grafting: insights from the TiCAB trial. Eur J Cardiothorac Surg. 2020 Apr 1;57(4):732-739. doi: 10.1093/ejcts/ezz313. PMID 31750899
- [Derived] Schunkert H, Boening A, von Scheidt M, Lanig C, Gusmini F, de Waha A, Kuna C, Fach A, Grothusen C, Oberhoffer M, Knosalla C, Walther T, Danner BC, Misfeld M, Zeymer U, Wimmer-Greinecker G, Siepe M, Grubitzsch H, Joost A, Schaefer A, Conradi L, Cremer J, Hamm C, Lange R, Radke PW, Schulz R, Laufer G, Grieshaber P, Pader P, Attmann T, Schmoeckel M, Meyer A, Ziegelhoffer T, Hambrecht R, Kastrati A, Sandner SE. Randomized trial of ticagrelor vs. aspirin in patients after coronary artery bypass grafting: the TiCAB trial. Eur Heart J. 2019 Aug 1;40(29):2432-2440. doi: 10.1093/eurheartj/ehz185. PMID 31145798